CLINICAL TRIAL: NCT01613521
Title: Tumor Perfusion and Hypoxia Assessed by DCE-MRI and 18F-FMISO PET as Biomarkers of Treatment Response in Cervical Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-174
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Cervical Cancer
Keywords: DCE-MRI; 18F-FMISO PET; 11-174
MeSH Terms: conditions — Uterine Cervical Neoplasms

ARMS (1):
- DCE-MRI and 18F-FMISO PET (Experimental): Each patient will undergo three DCE-MRI (dynamic contrast-enhanced MRI) studies: a baseline DCE-MRI within two weeks before chemoradiation; a second DCE-MRI after the second week of treatment (within a week); and a third DCE-MRI three months after treatment. As a pilot study in 10 patients, we will perform 18F-FMISO PET/CT on the same day of a baseline DCE-MRI before chemoradiation. Treatment decisions will not be based on DCE-MRI and 18F-FMISO PET/CT studies.
  Interventions: Other: DCE-MRI and 18F-FMISO PET

INTERVENTIONS:
Other: DCE-MRI and 18F-FMISO PET — DCE-MRIs: (i) Baseline DCE-MRI within two weeks before chemoradiation; (ii) Second DCE-MRI after the second week of chemoradiation (within a week); (iii) Third DCE-MRI three months after chemoradiation. iii. 18F-FMISO PET: Baseline 18F-FMISO PET within two weeks before chemoradiation (only 10 patients as a pilot study). iv. Clinical Follow-up: (i) Physical examination (every 3 months); (ii) Pap smear or cervical biopsy (every 3 months); (iii) follow-up imaging studies (CT and/or MRI) as per routine clinical follow-up of patients.

SUMMARY:
This study is to assess how patients respond to their treatment for cervical cancer. This research does not involve a specific treatment for the cancer that will be recommended by the doctor and may include radiation therapy and/or chemotherapy. This is a separate research imaging study designed to assess how patients respond to their treatment for cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-documented, newly-diagnosed primary cervical cancer of all histopathology types.
* Clinically visible gross lesion (International Federation of Gynecology and Obstetrics (FIGO) stage IB1 and above).
* Treatment (chemoradiation), DCE-MRI and 18F-FMISO PET studies will be at MSKCC.
* Patients must be an adult female 18 years of age or older.

Exclusion Criteria:

* Patients who because of general medical or psychiatric condition, or physiologic status cannot give an informed consent.
* Patients who received prior radiation treatment to pelvis.
* Patients with contraindications to DCE-MRI (non-compatible cardiac pacemakers or intracranial vascular clips, allergy to Gadolinium, end-stage renal disease) and/or 18F-FMISO PET.
* Patients who do not fulfill the screening criteria for safe DCE-MRI or 18F-FMISO PET as per the Department of Radiology guidelines.
* Pregnant patients; and or patients who are breast-feeding their babies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
predict tumor response | 2 years
  For each DCE-MRI parameter, the relative percent change from baseline to the two-week measurement will be calculated. These values will be assessed using ROC curves to evaluate whether they are predictive of tumor response.

SECONDARY OUTCOMES:
predict disease-free survival | 2 years
  baseline tumor perfusion parameters are predictive of disease-free survival at 2 years and 5 years, the primary analysis will again be an ROC analysis, but with the ROC curves modified to take into account the censored failure-outcome. We will create time-dependent ROC curves using methods described by Heagerty et al.

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Akin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/cancer-care/doctor